CLINICAL TRIAL: NCT04895969
Title: Prevalence of Partial Edentulism Among Patients of Faculty of Dentistry Cairo University
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmien Emad Eldeen, resident at prosthodontics deparetment and Master student at prosthodontics deparetment., Cairo University
Other Study IDs: Prevalence
Record Dates: First submitted 2021-05-17; First posted 2021-05-21 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2022-03

CONDITIONS: Partial-edentulism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The patterns of tooth loss are evaluated in many selected populations in numerous countries and so the frequency of partial edentulism seems to vary widely between different countries.

The prevalence of various patterns of partially edentulous arches should be frequently revised and updated .

This could help identify the changing treatment needs of the population and provide guidelines to prevent tooth loss emphasis should be placed on dental education, improve the quality of prosthodontic care being provided to patients oral and general health promotion which should highlight the control of common oral diseases such as caries at their various stages of progression and periodontal diseases.

Additionally, regular dental check-ups should be made mandatory at schools, colleges and workplaces and community field trips should be conducted in order that increase in oral health awareness can also discourage patients attitude waiting until acute symptoms develop.

According to our knowledge, no available studies investigated the prevalence of partial edentulism among patients in faculty of dentistry Cairo university. Therefore, this study wouldbe of valuable information to oral health planners for proposing strategies that will help dentalhealth care management in faculty of dentistry Cairo,

DETAILED DESCRIPTION:
study will be conducted on Patients above age of 20 years irrespective of sex, race, socioeconomic status having partially edentulism in either or both the arches to detect incidence and occurence of partial edentlism then detect its prevalance

ELIGIBILITY:
Inclusion Criteria:

* Study population who satisfied following criteria were included in the study:

  1. Patients above age of 20 years irrespective of sex, race, socioeconomic status having partially edentulism in either or both the arches
  2. Individuals who are willing and cooperative for study

Exclusion Criteria:

1. Completely edentulous patients,
2. patients with teeth extracted for orthodontic purpose
3. Patients with an only missing third molar, un erupted or congenitally missing teeth, root tips,and loose teeth that were indicated for extraction were not included in the study.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Partially edentulous patients of unknown classes
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Different Kennedy classes | "through study completion, an average of 1 year"
  Prevalence of partial edentulism among patients of Faculty of Dentistry Cairo University

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1.Muneeb, A., Khan, B. M., & Jamil, B. (2013). Causes and pattern of partial edentulism/exodontia and its association with age and gender: semi rural population, Baqai Dental college, Karachi, Pakistan. International Dental Journal of students research, 1, 13-18. 2.Sapkota, B., Adhikari, B., & Upadhaya, C. (2013). A Study of Assessment of Partial edentulous patients based on Kennedy's classification at Dhulikhel Hospital Kathmandu University Hospital. Kathmandu University Medical Journal, 11(4), 325-327. 3. Bharathi, M., Babu, K. R., Reddy, G., Gupta, N., Misuriya, A., & Vinod, V. (2014). Partial Edentulism based on Kennedy's classifcation: an epidemiological study. The journal of contemporary dental practice, 15(2), 229- 231. 4. Madhankumar, S., Mohamed, K., Natarajan, S., Kumar, V. A., Athiban, I., & Padmanabhan, T. V. (2015). Prevalence of partial edentulousness among the patients reporting to the Department of Prosthodontics Sri Ramachandra University Chennai, India: An epidemiological study. Journal of pharmacy & bioallied sciences, 7(Suppl 2), S643. 5. Nayyer, M., Khan, D. A., Gul, H., Aslam, A., Khan, N. B., & Aslam, F. (2020). Patterns of partial edentulism according to kennedy's classification-a cross sectional study. Pakistan Armed Forces Medical Journal, 70(Suppl-1), S87-90. 6. World Health Organization. Oral Health Surveys: Basic Methods, 4th ed. Geneva: WHO; 2014.